CLINICAL TRIAL: NCT04947943
Title: Impact of Geriatric Care in the Treatment of Older People Hospitalised for COVID-19
Brief Title: Geriatric Care for Older People Hospitalised for COVID-19
Acronym: COVAGERT
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0372
Record Dates: First submitted 2021-06-30; First posted 2021-07-01 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Covid19
Keywords: COVID-19; Comprehensive geriatric assessment (CGA); Older adults
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — myocardial fragments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Current COVID-19 pandemic implies regular treatment adaptation by physician, according to scientific publication evolution. Older adults are particularly affected by COVID-19, with the higher severe form prevalence and the higher mortality rate. Furthermore older peoples are at high risk of complications cascade, due to the SARS-Voc-2 infection but also because of chronic diseases decompensation. If risk factors in this population have been identified, specific treatments to reduce complications or to be curative are less known. However geriatric care, thanks to its holistic approach, could reduce these complications and improve survival.

Our study aims to determine if geriatric care provided in geriatric COVID-19 hospitalisation units improves survival of older people (aged 65 years and over) at one month in comparison with conventional COVID-19 hospitalisation unit during the first wave in the Montpellier University Hospital. Secondary objectives are to determine if clinical characteristics of older patients are different between conventional and geriatric COVID-19 hospitalisation units, to assess influence of clinical characteristics of older patients on their survival, and to determine wich treatment have been delivered for older people during the COVID-19 pandemic first wave in our hospital in view of bibliographic data available at this time.

COVAGERT is a monocentric, descriptive, observational and retrospective study, including all older adults aged 65 years and over hospitalised in the geriatric COVID-19 and the conventional COVID-19 units of the Montpellier University Hospital during the first wave of the SARS-Cov-2 pandemic (between March 1th 2020 and September 1th 2020). Principal outcome is the survival one months after the RT-PCR positive test. Some data about treatments, medical history, socio-demographic and clinical characteristics will be collected from the medical record.

Statistical analysis will be performed using univariate and multivariate regressions according to the study's objectives.

Results will be useful to determine the bring of geriatric care during the current pandemic, but also to highlight the importance of multidisciplinary assessment in this complex disease and for further emergency medical challenges.

ELIGIBILITY:
Inclusion criteria:

* adult age 65 years or over
* hospitalised for COVID-19 in one of the two hospitalisation unit (conventional or geriatric) during the first COVID19 wave

Exclusion criteria:

- refusal to give the access to her/his medical record

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older adults aged 65 years and over, hospitalised in the conventional or the geriatric COVID-19 hospitalisation unit during the first COVID-19 wave in the Montpellier University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
survival one month after positive SARS Cov 2 RT-PCR test | day 1
  survival one month after positive SARS Cov 2 RT-PCR test

SECONDARY OUTCOMES:
number of delivered treatments | day 1
  delivered treatments
type of clinical characteristics | day 1
  type of clinical characteristics
type of socio-demographic characteristics | day 1
  type of socio-demographic characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Miot stéphanie, PH, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC